CLINICAL TRIAL: NCT04220281
Title: Comparison of the Hypotensive Efficacy of Propofol Infusion Versus Nitroglycerin Infusion in Functional Endoscopic Sinus Surgery
Brief Title: Comparison Between Two Drugs (Propofol and Nitroglycerin as a Hypotensive Agents During Endoscopic Sinus Surgery
Acronym: prop
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: the number of patients needed for the study have been collected
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rasha Gamal Abusinna, lecturer of anesthesia and intensive care, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RGAbusinna
Record Dates: First submitted 2020-01-04; First posted 2020-01-07 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Hypotensive Anesthesia
Keywords: propofol; nitroglycerin
MeSH Terms: interventions — Propofol; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol group (Active Comparator): propofol group will receive propofol infusion
  Interventions: Drug: Propofol
- nitroglycerin group (Active Comparator): will receive nitroglycerin infusion
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Propofol — propofol infusion during surgery
  Other Names: prop
  Arms: propofol group
Drug: Nitroglycerin — nitroglycerin infusion during surgery
  Other Names: NTG
  Arms: nitroglycerin group

SUMMARY:
Background and Objectives: FESS is a common minimally invasive surgery that requires a clear field to be performed well. Hypotensive anesthesia is one of the most common maneuvers performed to help in keeping the field clear. An ideal drug for hypotensive anesthesia should be cheap and familial to the anesthesiologist. So being familial with propofol and by using its cardio-depressant action the idea of the research was developed and comparing it with nitroglycerin (a hypotensive agent in our protocol). Methods: The patients agreed to participate in the research were classified into two groups for comparison. Propofol group; received propofol infusion all over the procedure, and nitroglycerin group; received nitroglycerin infusion all over the procedure. Duration of surgery, visibility of surgical field and amount of blood loss were recorded. Pulse/min and MAP were recorded at baseline and every 5 min. Results: The mean duration of surgery was longer in the NTG to propofol group. There was high statistical significance in the average blood loss in the propofol group compared to NTG group. The visibility of the operative field also was significant in the propofol group as compared to NTG group. The mean heart rate in the NTG group is higher than the mean heart rate in the propofol group. The MAP in both groups is within a close range. Conclusion: Propofol and NTG can produce a safe and effective controlled hypotension during FESS. Whereas, propofol has; a better surgical field visibility, less surgical bleeding and less tachycardia during FESS.

DETAILED DESCRIPTION:
1. INTRODUCTION FESS (functional endoscopic sinus surgery) is a popular minimally invasive surgical technique for management of patient with sinus pathological conditions. The aim of this sinus endoscopic surgery is to restore a normal mucociliary clearing function and drainage of sinuses. Although, it is a minimally invasive surgery but it can lead to a serious complications such as optic nerve injury, orbital cellulitis, meningitis, and rhino-oral fistulas. Bleeding is one of the obstacles that is associated with this technique that can decrease the surgical field visualization and increase the probability of complications.

   One of the most important maneuvers used to minimize this bleeding is hypotensive anesthesia. The ideal hypotensive agent for anesthetist must be a familiar drug, easy to use, rapid onset and offset and with minimal side effects. Nitroglycerin infusion is a frequently used drug to produce controlled hypotension, as it is cheap and easy to use drug rapid onset and offset time. But a common side effect is reflex tachycardia and venous congestion which may also obscures the surgical filed and decreases surgeon satisfaction.

   Total intravenous anesthesia (TIVA) using propofol and remifentanil is a common procedure used in western countries. In Egypt remifentanil is not freely available. So this study will be designed to use inhalational anesthesia and use propofol infusion as a hypotensive agent and to determine whether controlled hypotension, surgeon's satisfaction and better operative filed can be achieved when compared to nitroglycerine infusion.
2. AIM OF THE WORK The aim of the study is to identify the efficacy of propofol infusion as a hypotensive agent in comparison with nitroglycerin infusion during FESS.

Study Design

A total of 40 adult patients undergoing FESS procedure for sinusitis. Written informed consent will be obtained from all patients before randomization. Patients will be divided equally into two groups the first 20 patients will be assigned to propofol group (Prop group) and the other group to nitroglycerin group (NTG group). Group assignment, preparation and administration of drugs will be performed by a junior anesthetist who is neither involved nor interested by any means in the study. The patients, the ENT surgeon, and the anesthetist collecting data all were blind to the groups. The anesthetist performing the general anesthesia was not blinded to the drug given but he was not one of the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA I and II diagnosed for chronic sinusitis
* Age range between 18-60 years, undergoing elective FESS without septoplasty under general anesthesia.

Exclusion Criteria:

* included any patient with bleeding disorder, on anticoagulant therapy
* renal, hepatic or cardiac dysfunction
* history of cerebrovascular stroke
* peripheral vascular diseases
* allergic to any of the study drugs
* hypertension
* morbid obesity and
* recurrent endoscopic sinus surgeries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
efficacy of propofol infusion as a hypotensive agent in comparison with nitroglycerin infusion in FESS surgeries under general anesthesia | the study data collected during the time of surgery ranging from 1-2 hours
  measuring MAP every 5 min all over the time of surgery comparing the two study groups (propofol infusion versus nitroglycerin infusion)

SECONDARY OUTCOMES:
measuring the pulse rate | the study data collected during the time of surgery ranging from 1-2 hours
  comparing the pulse rate (beat/min) every 5 min all over the time of surgery comparing the two study groups (propofol infusion versus nitroglycerin infusion)
visibility of the surgical field by using the Average Category Scale | done by the surgeon immediately after the surgery
  evaluation of the visibility of the operative field during surgery by using the average category scale. minimum is grade 0 and maximum grade 5. the less the grade the better the visibility of the surgical field.
amount of blood loss | done by the anesthetist every 1 hour during the surgery
  measuring the amount of blood lost during the surgery by ml/hr

CONTACTS AND LOCATIONS:
Overall Officials: Rasha G Abusinna, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, EL Abassia, Egypt